CLINICAL TRIAL: NCT01303874
Title: A Multicentre Randomised Trial Of Etanercept And Methotrexate To Induce Remission In Early Inflammatory Arthritis
Brief Title: Etanercept and Methotrexate in Patients to Induce Remission in Early Arthritis (EMPIRE)
Acronym: EMPIRE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Paul Emery, Professor, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RR05/7150; 2005-005467-29 (EudraCT Number)
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Rheumatoid Arthritis; Inflammatory Arthritis
Keywords: Rheumatoid arthritis; Inflammatory arthritis; Undifferentiated arthritis; Etanercept; Combination Therapy
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Etanercept; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination Therapy (Experimental): Methotrexate & Etanercept
  Interventions: Drug: Etanercept (ETN)
- Single-agent therapy (Placebo Comparator): Methotrexate (MTX)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etanercept (ETN) — ETN 50 mg subcutaneous (SC) injections once weekly and MTX orally once weekly.
  Other Names: Enbrel
  Arms: Combination Therapy
Drug: Placebo — ETN-matching placebo SC injections once weekly and MTX orally once weekly.
  Other Names: Maxtrex
  Arms: Single-agent therapy

SUMMARY:
TRIAL DESIGN

1. Description This is a 18-month, double-blind, randomized, multicentre, outpatient study. The approximate duration of subject participation will be 18 months and the approximate total duration of the study will be 42 months. The duration of subject enrollment will be approximately 24 months.
2. Discussion of Trial Design The study is designed to directly compare the effectiveness of combination therapy with MTX + ETN versus
3. Principal research question/objective To determine the number of patients in clinical remission at 12 months of follow-up, as defined as the absence of symptoms and signs of inflammatory arthritis.

DETAILED DESCRIPTION:
Early arthritis is frequently undifferentiated. It is well recognised that a substantial proportion of patients with an undifferentiated inflammatory arthritis will go on to develop persistent synovitis, with the strongest predictor of persistence being disease duration > 12 weeks (1-4). Studies have shown that patients with early oligoarthritis who fail to respond within 2 weeks to corticosteroid injections have a high likelihood of persistent disease (2). It is therefore clear that these patients with early inflammatory arthritis need definitive treatment, but the optimal therapeutic strategy is yet to be determined.

Tumor Necrosis Factor (TNF) is a naturally occurring cytokine that is involved in normal inflammatory and immune responses. It plays an important role in the inflammatory process of rheumatoid and other arthritis, and the resulting joint pathology. Elevated levels of TNF are found in the synovial fluid of patients with RA. Two distinct receptors for TNF exist naturally as monomeric molecules on the cell surfaces and in soluble forms. Biological activity of TNF is dependent upon binding to either cell surface TNF receptors (TNFR). Etanercept (ETN) is a dimeric fusion protein consisting of the p75 TNFR linked to the Fc portion of human IgG1, and is capable of binding two TNF molecules. Etanercept inhibits binding of both TNF-alpha and TNF-beta to cell surface TNFRs, rendering TNF biologically inactive. Agents that block TNF are effective in all types of arthritis (with the exclusion of connective tissue diseases).

It is generally agreed that there is a window of opportunity in active early inflammatory arthritis in which definitive treatment may give a disproportionate improvement compared to treatment at a later time, and may well be able to induce remission in a subgroup of patients.

Studies in early rheumatoid arthritis (< 12 months) have shown that remission-induction with the TNF-antagonist infliximab provides a significant reduction in MRI-evidence of synovitis and erosions at 12 months with evidence of sustained functional and quality of life benefits at 2 years, despite withdrawal of infliximab at 12 months (5). Results from the TEMPO study show that treatment of established rheumatoid arthritis with ETN+MTX achieves remission in about 40% patients (6). TNF antagonists also have the therapeutic benefit of rapid and sustained suppression of inflammation.

Treatment of patients with early undifferentiated arthritis with ETN+MTX is hypothesised to prevent progression of persistent disabling disease in a significant number of patients. Induction of remission at this time in the disease course may result in sustained remission, reduce the need for further treatment, and be most cost effective therapeutic strategy.

ELIGIBILITY:
Inclusion Criteria:

* Is age 18 -80 years old
* Patients have articular synovitis, within 3 months of diagnosis
* Either RF antibody (+) or anti-CCP antibody (+) or SE (+)
* Demonstrates a negative urine pregnancy test at screening if female of childbearing potential
* Agrees to use a medically accepted form of contraception during the study and for 3 months after the last dose of study drug, if sexually active male
* Is capable of understanding and signing an informed consent form
* Is able and willing to self-inject study drug or have a designee who can do so
* Is able and willing to take oral medication
* Is able to store injectable test article at 2° C to 8° C
* Demonstrates a negative tuberculosis screening test

Exclusion Criteria:

* Received previous treatment with any DMARDS
* Received previous treatment with ETN or other tumour necrosis factor (TNF) antagonist (e.g. a TNF monoclonal antibody or a soluble TNF-receptor)
* Previous treatment with IL-1 receptor antagonist
* Chronic arthritis diagnosed before 16 years old
* Received any investigational "biological" agent within 3 months of screening visit
* Received treatment with any investigational drug of "chemical" nature within one month prior to study screening
* Known Human Immunodeficiency Virus (HIV)
* Presence of any contraindication to ETN or MTX
* Has significant concurrent medical diseases
* Has cancer or a history of cancer within 5 years of entering the screening period
* Current crystal or infective arthritis
* Chronic infection of the upper respiratory tract, chest, urinary tract or skin
* Any ongoing or active infection or any major episode of infection requiring hospitalization or treatment with IV antibiotics within the preceding 30 days and/or orally administered antibiotics in the preceding 15 days
* Demonstrates liver function abnormality
* Has renal disease
* Has leukopenia
* Has thrombocytopenia
* Has a hemoglobin level of < 9g/L for males and < 85 g/L for females
* Is pregnant or breast-feeding
* Joint surgery within preceding 2 months (at joints to be assessed within this study)
* Received anti-CD4, diphtheria interleukin-2 fusion protein, anti-interleukin-6 (anti-IL-6), rituximab or other immunosuppressive biologic during the last 6 months before screening, and treatment with such agents more than 6 months before screening if there are persistent signs of immunosuppression (with a subsequent abnormal absolute T-cell count) at screening visit
* Received any live (attenuated) vaccines within 4 weeks of screening visit
* Received cyclophosphamide within 6 months of screening visit
* Any corticosteroids within 28days prior to screening
* Uses a dose of NSAID greater than the maximum recommended dose in the product information at the screening visit
* Has a history of confirmed blood dyscrasia
* Has any condition judged by the physician to cause this study to be detrimental to the subject
* Has a history of drug abuse or psychiatric disease that would interfere with the ability to comply with the study protocol
* Has a history of alcohol abuse or excessive alcohol beverage consumption
* Has a history of known liver cirrhosis, fibrosis, or fatty liver
* Has a history of any viral hepatitis within 1 year of screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2006-09; Primary Completion 2010-11-05 (Actual); Study Completion 2010-11-05 (Actual)

PRIMARY OUTCOMES:
clinical remission | 12 months
  To determine the number of patients in clinical remission at 12 months, as defined as the absence of symptoms and signs of inflammatory arthritis (i.e. swollen joint count 0; tender joint count 0)

SECONDARY OUTCOMES:
clinical remission | 18 months
  The number of patients in clinical remission at 18 months (as defined as absence of symptoms and signs of clinical arthritis i.e. swollen joint count 0 ; tender joint count 0)
Conventional disease activity measures | week 78
  Conventional disease activity measures (VAS pain/fatigue/global/physician, EMS, TJC, SJC, CRP, ESR)
Functional, work and quality of life assessments | Week 78
  Functional, work and quality of life assessments (HAQ, WIS, WDA, EQ-5d, SF-36)
remission | Week 26
  Proportion of patients achieving 26 weeks of remission
DAS 44 | Week 78
  Disease Activity Score (DAS) 44
drug-free remission | 12 & 18 mths
  The number of patients in drug-free remission at 12 18 months
etanercept-free remission | 12 and 18 months
  The number of patients in etanercept-free remission at 12 and 18 months (ETN arm)
Remission by ACR Criteria | Week 78
  Remission by ACR Criteria
effects of the combination of ETN and MTX to MTX alone on radiographic change | 12 months and 18 months
  To compare the effects of the combination of ETN and MTX to MTX alone on radiographic change at 12 months and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Emery, Prof, Principal Investigator — University of Leeds
Locations (1):
- Leeds Teaching Hospital HNS Trust, Leeds, West Yorkshire, United Kingdom